CLINICAL TRIAL: NCT03294941
Title: The HepQuant SHUNT Test for Monitoring Liver Disease and Treatment Effects by Measuring Liver Function and Physiology
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Primary study stopped early
Sponsor: HepQuant, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: HQ-US-SHUNT-1701
Record Dates: First submitted 2017-03-30; First posted 2017-09-27 (Actual); Results first posted 2021-07-15 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: All subjects receive HepQuant SHUNT test and DSI measurement, but must first be enrolled into one of the three Gilead clinical trials listed above before they can be enrolled in the HepQuant study. Since the assigned intervention, the HepQuant SHUNT test, is the same for all participants in all three Gilead clinical trials, there is only one arm and intervention for the HepQuant study itself. Some analyses are conducted by grouping subjects into those who took the placebo in the parallel drug study versus those who were on active study drug in the parallel study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- HepQuant SHUNT Liver Diagnostic Kit (Other): All subjects receive HepQuant SHUNT test and DSI measurement. HepQuant SHUNT is a combination product where 13C Cholate 20mg is administered intravenously once for each test and d4 Cholate 40mg is administered once orally for each test
  Interventions: Combination Product: HepQuant SHUNT Liver Diagnostic Kit

INTERVENTIONS:
Combination Product: HepQuant SHUNT Liver Diagnostic Kit — Serial testing over 48 weeks
  Other Names: SHUNT test

SUMMARY:
The HepQuant SHUNT test, which is provided as a HepQuant SHUNT Liver Diagnostic Kit, is a minimally-invasive test of liver function and physiology which has been designated by the FDA as an investigational drug/device combination product.

Enrollment into one of the 3 Gilead Selonsertib clinical trials (GS-US-416-2124, GS-US-384-1943/1944) is required for enrollment into the HepQuant study

DETAILED DESCRIPTION:
The HepQuant study is to run parallel to the Gilead clinical trials,GS-US-416-2124 trial of Alcoholic Hepatitis, GS-US-384-1943 trial of non-alcoholic steatohepatitis (NASH) fibrosis Stage 3 (STELLAR-3), and, GS-US-384-1944 trial of NASH and compensated cirrhosis (STELLAR-4). The time points for the HepQuant SHUNT tests coincide with pre-specified time points within the Gilead clinical trials. Subjects enrolled in GILEAD's STELLAR and Alcoholic hepatitis trials may participate concurrently in this HepQuant sponsored investigational device study at participating US sites only (IDEs as listed above) once approved by the applicable IRB/IEC.

The main eligibility criteria for enrollment into the HepQuant study is enrollment into one of the three Gilead clinical trials listed above.

The HepQuant SHUNT Test is minimally-invasive and measures hepatocyte function and inflow to the liver from the simultaneous clearances (hepatic filtration rates, HFRs) of cholate from systemic and portal circulations. The Test quantifies portal-systemic shunting (SHUNT) and generates a liver disease severity index (DSI). DSI is a score from 0 (no disease) to 50 (terminal illness) that is a composite of both HFRs and correlates with stage of fibrosis, presence of varices, especially large varices, and risk for future clinical outcomes. DSI is the primary output variable from the HepQuant SHUNT test. The HepQuant SHUNT test potentially satisfies the unmet medical need for a minimally-invasive test of global liver function and physiology

ELIGIBILITY:
Inclusion Criteria:

The key inclusion criteria for this HepQuant Parallel Study are the inclusion criteria into one of the Gilead selonsertib trials (GS-US-416-2124, GS-US-384-1943 or 1944). Once that has been met, subjects must:

* Be able to ingest liquid by mouth
* Have venous access to support a peripheral IV and 6 blood draws

Exclusion Criteria:

The key exclusion criteria for this HepQuant Parallel Study are the exclusion criteria for one of the Gilead selonsertib trials (GS-US-416-2124, GS-US-384-1943 or 1944). If this has been met, the subject is not eligible to participate in HepQuant. If no exclusion criteria has been met for the Gilead selonsertib trial, ADDITIONAL exclusions for HepQuant are:

* Subject should not have had first dose of selonsertib
* Subject cannot take anything by mouth
* Subject cannot be hypersensitive to eggs, albumin preparations, any ingredient in the formulation, or component of the container
* Subject cannot have intercurrent medical or surgical illness (eg: acute MI, acute cerebral hemorrhage, sepsis)
* subject cannot have had extensive resection of large segments of small intestine (short gut)
* Subject cannot have severe gastroparesis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2019-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greg Everson, MD, Study Director — HepQuant, LLC
Locations (8):
- United States (8):
  - Schiff Center for Liver Diseases, Miami, Florida
  - University of PA, Philadelphia, Pennsylvania
  - Methodist Dallas Medical Center, Dallas, Texas
  - TX Digestive Disease Consultants, Dallas, Texas
  - The Texas Liver Institute, San Antonio, Texas
  - McGuire VA Med Cntr, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washingtion, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- HepQuant SHUNT Liver Diagnostic Kit - Placebo in Parallel Study; HepQuant SHUNT Liver Diagnostic Kit - Active Study Drug in Parallel Study: All subjects receive HepQuant SHUNT test and DSI measurement. HepQuant SHUNT is a combination product where 13C Cholate 20mg is administered intravenously once for each test and d4 Cholate 40mg is administered once orally for each test
  HepQuant SHUNT Liver Diagnostic Kit: Serial testing over 48 weeks
Period: Overall Study
Arm/Group | HepQuant SHUNT Liver Diagnostic Kit - Placebo in Parallel Study | HepQuant SHUNT Liver Diagnostic Kit - Active Study Drug in Parallel Study
Started | 4 | 13
Completed | 4 | 11
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HepQuant SHUNT Liver Diagnostic Kit - Placebo in Parallel Study | HepQuant SHUNT Liver Diagnostic Kit - Active Study Drug in Parallel Study | Total
Number analyzed (Participants) | 4 | 13 | 17
Age, Continuous [Mean (Full Range); unit: years] | 48.75 [28 to 57] | 58.15 [44 to 69] | 55.94 [28 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 11 | 15
  Male | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 7 | 10
  Not Hispanic or Latino | 1 | 6 | 7
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 13 | 17

OUTCOME MEASURES:

1. Primary Outcome: Baseline DSI
Description: The baseline DSI, or disease severity index, is a measure of severity of liver disease at baseline. The scores for DSI range on a scale from 0 (healthy liver) to 50 (severe liver disease).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HepQuant SHUNT Liver Diagnostic Kit - Placebo in Parallel Study | HepQuant SHUNT Liver Diagnostic Kit - Active Study Drug in Parallel Study
Number analyzed (Participants) | 4 | 13
score on a scale | 21.63 (3.31) | 20.93 (3.55)

2. Primary Outcome: Change in DSI From Baseline to 48 Weeks
Description: Improvement or worsening of liver disease severity from baseline to the week 48 visit as measured by the change in the disease severity index (DSI) (DSI at 48 weeks minus DSI at baseline). The scores for DSI range on a scale from 0 (healthy liver) to 50 (severe liver disease).
Time Frame: Baseline and at 48 weeks
Population: 15 subjects completed the week 48 SHUNT Test (4 in parallel study placebo group, and 11 in parallel study active study drug group), however, the SHUNT Test samples were unanalyzable for 1 subject on active study drug due to failure of the IV Clearance component of the SHUNT Test. Therefore, the present analysis only includes 14 subjects (4 on placebo, 10 on active study drug).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HepQuant SHUNT Liver Diagnostic Kit - Placebo in Parallel Study | HepQuant SHUNT Liver Diagnostic Kit - Active Study Drug in Parallel Study
Number analyzed (Participants) | 4 | 10
score on a scale | -1.08 (2.44) | -1.00 (2.28)

3. Secondary Outcome: Severity of Liver Disease Index (DSI) Scores Stratified by Baseline NASH CRN Stage of Fibrosis
Description: Compared baseline disease severity index (DSI) scores, which are used to measure severity of liver disease on a scale from 0 (healthy liver) to 50 (severe liver disease), between subjects with F3 or F4 Fibrosis at baseline. Fibrosis stages were obtained clinically using the NASH CRN Scoring System to grade liver biopsy results. This scoring system yields scores ranging from F0 (no fibrosis/healthiest) to F4 (cirrhosis/severe disease). Subjects in this study either had F3 Fibrosis (bridging fibrosis) or F4 Fibrosis (cirrhosis), so F3 subjects have less severe disease than F4 subjects.
Time Frame: Baseline
Population: Analysis was conducted to compare DSI scores between Fibrosis categories instead of by placebo vs active study drug groups because the subject numbers were too low. There was only one subject in the placebo group with F4 Fibrosis. Additionally, this outcome measure was established to compare DSI scores to other liver disease severity scores regardless of study drug use, so this analysis was conducted by grouping fibrosis scores.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- HepQuant SHUNT Liver Diagnostic Kit - Subjects With F3 Fibrosis; HepQuant SHUNT Liver Diagnostic Kit - Subjects With F4 Fibrosis: All subjects receive HepQuant SHUNT test and DSI measurement. HepQuant SHUNT is a combination product where 13C Cholate 20mg is administered intravenously once for each test and d4 Cholate 40mg is administered once orally for each test
  HepQuant SHUNT Liver Diagnostic Kit: Serial testing over 48 weeks
Arm/Group | HepQuant SHUNT Liver Diagnostic Kit - Subjects With F3 Fibrosis | HepQuant SHUNT Liver Diagnostic Kit - Subjects With F4 Fibrosis
Number analyzed (Participants) | 9 | 8
score on a scale | 19.39 (1.70) | 23.02 (3.91)

ADVERSE EVENTS:
Time Frame: 12 months, from the date of enrollment through the 48 week/final study visit.
Description: Adverse events are all grouped together because the only intervention in the HepQuant Study is the HepQuant SHUNT Test. Although some analyses are conducted by grouping subjects into those who took the placebo in the parallel drug study versus those who were on active study drug in the parallel study, the HepQuant study itself had only one arm.
Arm/Group | HepQuant SHUNT Liver Diagnostic Kit
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 3/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HepQuant SHUNT Liver Diagnostic Kit (N=17)
Mild IV-related events (Injury, poisoning and procedural complications) | 3 (3) — Mild pain due to IV insertion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/41/NCT03294941/Prot_SAP_000.pdf